CLINICAL TRIAL: NCT04776733
Title: Comparing the Efficacy and Tolerability of a Prepackaged Semisolid Nutritional Formulations With a Restricted Diet for Colonoscopy Preparation: A Randomized Clinical Trial.
Brief Title: Prepackaged Nutritional Formulations Versus Restricted Diet for Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: AHE 1.0
Record Dates: First submitted 2021-02-24; First posted 2021-03-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prepackaged group (Experimental): All colonoscopy were performed in the afternoon. The day before the colonoscopy: 3 bags of pre-packaged food were used for diet preparation. All the patients drink single dose of 60g Polyethylene Glycol (PEG-4000) with 1L water at a rate of 250 ml every 15 min in the evening.
  On the day of the colonoscopy: a bag of pre-packaged food were used for breakfast. All the patients drink single dose of 120g Polyethylene Glycol (PEG-4000) with 2L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Other: prepackaged semisolid nutritional formulations
- restricted diet group (Active Comparator): All colonoscopy were performed in the afternoon. The day before the colonoscopy: restricted diet prepared by patients were used for diet preparation. All the patients drink single dose of 60g Polyethylene Glycol (PEG-4000) with 1L water at a rate of 250 ml every 15 min in the evening.
  On the day of the colonoscopy: restricted diet prepared by patients were used for breakfast. All the patients drink single dose of 120g Polyethylene Glycol (PEG-4000) with 2L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Other: restricted diet

INTERVENTIONS:
Other: prepackaged semisolid nutritional formulations — The day before the colonoscopy: 3 bags of pre-packaged food were used for diet preparation.
  On the day of the colonoscopy: a bag of pre-packaged food were used for breakfast.
  Arms: prepackaged group
Other: restricted diet — The day before the colonoscopy: restricted diet prepared by patients were used for diet preparation.
  On the day of the colonoscopy: restricted diet prepared by patients were used for breakfast.
  Arms: restricted diet group

SUMMARY:
In order to analyze the effectiveness and patient tolerance of the two bowel preparation regimens, the investigators will compare prepackaged semisolid nutritional formulations and restricted diet. The aim was to demonstrate that prepackaged semisolid nutritional formulations is not inferior in overall quality of intestinal preparation to restricted diet in subjects undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18-75 years old requiring colonoscopy and willing to participate in this study.

Exclusion Criteria:

1. Patients with constipation;
2. Patients with congestive heart failure;
3. Patients with a history of kidney disease;
4. Patients with a history of poor intestinal preparation;
5. Pregnant / lactating women;
6. Patients without informed consent;
7. Allergic or intolerant to any research drug;
8. Patients with severe gastrointestinal diseases, such as intestinal obstruction or perforation, active ulcerative colitis, toxic colitis and toxic megacolon;
9. Patients with a history of inflammatory bowel disease;
10. History of colorectal resection；
11. Patients with diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | 1 Day of colonoscopy
  The OBPS，a scoring system with scores between 0 and 14, where 0 is the best score，divides the colon into 3 segments (right, transverse and rectosigmoid colon); each is scored from 0-4 (0=excellent, If it is necessary to suction liquid stool to adequately see the colonic wall, a score of 2 (fair) is given; if it is necessary to wash and to suction, a score of 3 (poor) is given. The remaining scores fall into place around these anchors. ). A score 0-2 is added to indicate the total amount of luminal fluid.(0=The total amount of fluid in the colon is very small,1=a moderate volume of fluid overall in the colon,2=a large volume of fluid overall in the colon)

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China